CLINICAL TRIAL: NCT05939388
Title: Battlefield Auricular Acupressure (BAApress) for Emergency Department Observation Psychiatric Patients With Co-occurring Chronic and Acute Pain Management
Brief Title: Battlefield Auricular Acupressure (BAApress) Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00098172
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Pain
Keywords: auricular acupressure; pain management; acupressure seeds; acute pain; chronic pain
MeSH Terms: conditions — Pain; Agnosia; Acute Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Auricular Acupressure Pad Group (Experimental): All subjects who qualify and agree to be in the study will be given Auricular Acupressure using an acupressure pad containing acupressure seeds for 4 days in addition to their regular standard of care pain medication.
  Interventions: Device: Auricular Acupressure Pads

INTERVENTIONS:
Device: Auricular Acupressure Pads — Pads containing seeds that are placed on specific sites of the ear that are thought to help with pain.

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) acupressure applied to the outside of the ear (Auricular Acupressure), in addition to the standard of care medication regimen, will have on pain. This study is being done to assess whether acupressure in addition to prescribed pain medication may be of benefit in decreasing pain levels and improving overall wellbeing. This study will also evaluate the feasibility of routinely offering acupressure to patients having pain issues in addition to a psychiatric diagnosis.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility of Emergency Department nurse-initiated battlefield auricular acupressure as an adjunct to medication for pain management for psychiatric Emergency Department Observation patients.

The Battlefield Auricula Acupressure interventionists (nurse) will complete Auricular training modules and complete competency assessments and intervention assessments throughout the study. Study interventionist will include the possibility that a study participant may be part of a competency assessment and that their session may be recorded and securely uploaded to a server per Institutional Review Board (IRB) and institutional policies.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring admission to psychiatric emergency room who also have documented chronic or acute pain
* History of chronic or acute pain with or without opioid use disorder
* Expected length of stay at least 2-3 days at the time of recruitment
* Able to read and understand the informed consent form

Exclusion Criteria:

* Since this is a feasibility pilot, only English-speaking participants will be eligible.
* Cognitive impairment (Intellectual Disability Disorder or Dementia)
* Patients who have a legal guardian
* Participants with a history of skin disease (e.g., psoriasis) involving the ear, adhesive allergy, recent scar tissue on ear, or current abrasions or cuts on ear,
* Use of some types of hearing aids (obstructing the placement of beads)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Olshan-Perlmutter, PMHCNS-BC, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Auricular Acupressure Pad Group
Started | 11
Completed | 10
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.64 (14.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 3
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Pain and General Activity Scores (Visual Analogue Scale)
Description: Visual Analogue Scale (VAS) for Pain is marked by subject on a line that ranges from 0mm to 100mm. The study team will measure where the participant marks to the nearest mm which will provide a score. Higher scores denote higher pain with higher levels of activity.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 11
mm | 65 [51.8 to 78.2]

2. Primary Outcome: Patient Reported Pain and General Activity Scores (Visual Analogue Scale)
Description: as for outcome 1
Time Frame: Day 1
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 11
mm | 57.3 [41.0 to 73.5]

3. Primary Outcome: Patient Reported Pain and General Activity Scores (Visual Analogue Scale)
Description: as for outcome 1
Time Frame: Day 2
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 11
mm | 52.7 [33.3 to 72.1]

4. Primary Outcome: Patient Reported Pain and General Activity Scores (Visual Analogue Scale)
Description: as for outcome 1
Time Frame: Day 3
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 10
mm | 42.2 [19.3 to 65.1]

5. Primary Outcome: Pain Medication Usage
Description: Average milligram per day of a non-opioid analgesic.
Time Frame: Day 1
Measure: Mean (95% Confidence Interval); unit: milligrams
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 11
milligrams | 291 [16 to 566]

6. Primary Outcome: Pain Medication Usage
Description: Average milligram per day of a non-opioid analgesic.
Time Frame: Day 2
Measure: Mean (95% Confidence Interval); unit: milligrams
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 11
milligrams | 871 [318 to 1425]

7. Primary Outcome: Pain Medication Usage
Description: Average milligram per day of a non-opioid analgesic.
Time Frame: Day 3
Measure: Mean (95% Confidence Interval); unit: milligrams
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 10
milligrams | 780 [394 to 1167]

8. Secondary Outcome: Battlefield Auricular Acupressure (BAA) Press Question 1 - Count of Participants Somewhat Satisfied or Satisfied.
Description: Number responding to the following question will be recorded:
  1. "How satisfied were you with how your pain has been treated?" using the Likert scale to measure "Very satisfied =5, Satisfied=4, Somewhat satisfied = 3, Somewhat dissatisfied= 2, Dissatisfied 1, Very Dissatisfied 0." Range 0-5 with higher score indicating higher satisfaction.
Time Frame: Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 10
Participants
  Very dissatisfied | 0
  Dissatisfied | 0
  Somewhat dissatisfied | 0
  Somewhat satisfied | 6
  Satisfied | 4
  Very satisfied | 0

9. Secondary Outcome: Battlefield Auricular Acupressure (BAA) Press Question 2 - Count of Participants That Would Maybe Consider or Consider Intervention.
Description: Number responding to the following question will be recorded:
  Would you consider using auricular acupressure in the future for pain or if recommended by your nurse or physician? a. No, would not use again (Score of 0) b. Maybe (Score of 1), c. Yes, I would consider using in the future (Score of 2).
Time Frame: Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 10
Participants
  Yes, I would consider using in the future | 8
  Maybe | 2
  No, would not use again | 0

10. Secondary Outcome: BAA Press Placement Survey (Interventionists Only) - Mean Time of Acupressure Seed Placement
Description: The Interventionist (Acupressure nurse) will be asked to capture time related to completion of study tasks and other qualitative questions to assess overall feasibility. Time recorded in minutes.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 11
minutes | 11.5 (3.7)

11. Secondary Outcome: General Anxiety Disorder Scale (GAD-7)
Description: GAD-7 is a 7 item scale to identify Generalized Anxiety Disorder symptoms of evaluation. Patients are asked to rate anxiety symptoms on a scale of 0-3. Total score ranges from 0-21. Higher scores indicate increased severity of anxiety.
  7 item scale to identify Generalized Anxiety Disorder symptoms of evaluation. Patients are asked to rate anxiety symptoms on a scale of 0-3. Total score ranges from 0-21. Higher scores indicate increased severity of anxiety
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 11
score on a scale | 15.0 [10.8 to 19.2]

12. Secondary Outcome: General Anxiety Disorder Scale (GAD-7)
Description: as for outcome 11
Time Frame: Day 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 11
score on a scale | 9.7 [4.4 to 15.1]

13. Secondary Outcome: General Anxiety Disorder Scale (GAD-7)
Description: as for outcome 11
Time Frame: Day 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 11
score on a scale | 7.1 [3.4 to 10.9]

14. Secondary Outcome: General Anxiety Disorder Scale (GAD-7)
Description: as for outcome 11
Time Frame: Day 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Auricular Acupressure Pad Group
Number analyzed (Participants) | 10
score on a scale | 5.7 [2.5 to 9.0]

ADVERSE EVENTS:
Time Frame: Baseline through day 3.
Arm/Group | Auricular Acupressure Pad Group
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT05939388/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT05939388/ICF_000.pdf